CLINICAL TRIAL: NCT06772272
Title: Effect of Perioperative Roxadustat in Elective Lumbar Interbody Fusion Surgery: a Parallel-group, Open-label, Randomised Controlled Trial.
Brief Title: Effect of Perioperative Roxadustat in Elective Lumbar Interbody Fusion Surgery.
Acronym: PRELIFS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Min Yan, Head of Department of Anesthesiology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0037
Record Dates: First submitted 2024-09-22; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-09

CONDITIONS: Perioperative Anemia
Keywords: Anemia; Roxadustat; Transfusion; Surgery
MeSH Terms: conditions — Anemia | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roxadustat (Experimental): Participants in this group will receive Roxadustat, administered orally at a dose of 100mg three times per week for a total of three weeks. This treatment will begin two weeks prior to the scheduled lumbar interbody fusion surgery and continue for one week postoperatively. The aim is to evaluate whether Roxadustat reduces perioperative blood transfusion requirements and assess its safety during the perioperative period.
  Interventions: Drug: Roxadustat
- Control (No Intervention): Participants in this group will receive standard clinical care according to the hospital's guidelines without the administration of Roxadustat. This group serves as a comparator to evaluate the effectiveness of Roxadustat in reducing perioperative blood transfusions during elective lumbar interbody fusion surgery.

INTERVENTIONS:
Drug: Roxadustat — Roxadustat is an oral hypoxia-inducible factor prolyl-hydroxylase inhibitor (HIF-PHI) used to treat anemia. Participants in the Roxadustat group will receive 100mg of Roxadustat orally three times per week for three weeks (two weeks prior to surgery and one week post-surgery). The dosage may be adjusted based on hemoglobin levels during the perioperative period: if hemoglobin rises above 150g/L, the drug will be stopped; if hemoglobin increases by more than 20g/L from baseline but is still below 130g/L, the dosage will be reduced to 70mg; if hemoglobin drops by more than 20g/L from baseline, the dosage will be increased to 120mg.
  Other Names: FG-4592; Evrenzo
  Arms: Roxadustat

SUMMARY:
The goal of this clinical trial is to assess whether Roxadustat can reduce perioperative blood transfusions in patients with anemia undergoing elective lumbar interbody fusion surgery. It will also evaluate the safety of Roxadustat in this context. The main questions it aims to answer are:

* Does Roxadustat reduce the need for perioperative red blood cell transfusions?
* Is Roxadustat safe for use in patients during the perioperative period?

Researchers will compare Roxadustat to standard clinical care without Roxadustat to determine its effectiveness and safety.

Participants will:

* Take Roxadustat orally three times a week for three weeks (two weeks before surgery and one week post-surgery).
* Undergo regular blood tests and follow-up monitoring during the hospital stay and up to 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, no upper age limit, sex unrestricted.
* Scheduled for elective lumbar interbody fusion surgery.
* Diagnosed with anemia (Hemoglobin levels: male <130g/L, female <120g/L).
* Willing to participate and able to voluntarily sign an informed consent form.

Exclusion Criteria:

* Patients admitted on an emergency basis.
* Patients with moderate to severe anemia (Hemoglobin levels <90g/L).
* Patients already enrolled in another clinical study.
* Patients unable to comply with the study protocol due to cognitive or language barriers.
* Pregnant or breastfeeding women.
* Patients who have already received erythropoiesis-stimulating agents, iron supplements, or other treatments to increase hemoglobin levels.
* Patients with severe infections.
* Patients with a history of acute coronary syndrome, heart failure, or cerebrovascular events within the last 3 months.
* Any other medical condition that may pose a safety risk, confound efficacy or safety evaluations, or interfere with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
Perioperative RBC transfusion requirement | Discharge or within 4 weeks of hospitalization (whichever comes first)
  The incidence of the composite outcome of perioperative transfusion requirement (defined as the occurrence of one or more of the following events):
  * Red blood cell transfusion
  * Perioperative lowest hemoglobin level below 80 g/L

SECONDARY OUTCOMES:
Blood Transfusion Rate | Discharge or within 4 weeks of hospitalization (whichever comes first)
  The percentage of participants in each group requiring red blood cell transfusion during the perioperative period.
Volume of Blood Transfused | Discharge or within 4 weeks of hospitalization (whichever comes first)
  The total volume of red blood cells transfused in units per participant during the perioperative period.
Hemoglobin Levels at Different Time Points | Baseline, pre-surgery, during surgery, 1, 3, 5, and 28 days post-surgery, and at 1 month and 6 months follow-up.
  Hemoglobin levels will be measured at key time points to assess changes, including: at baseline (enrollment), pre-surgery, during surgery, at 1, 3, 5, 28 days post-surgery, and at 1 month and 6 months follow-up visits to monitor longer-term effects.
Ferritin and Anemia-Related Blood Tests | Baseline, pre-surgery, 1, 3, 5, 28 days post-surgery.
  Levels of ferritin and other biomarkers related to anemia will be measured, including iron, transferrin, and vitamin B12, to assess the impact of Roxadustat on anemia.
Length of Hospital Stay | Discharge or within 4 weeks of hospitalization (whichever comes first)
  The total duration of hospitalization for each participant, measured in days.
Hospitalization Costs | Discharge or within 4 weeks of hospitalization (whichever comes first)
  The total cost of the hospital stay for each participant, including all treatments and care.
Thrombotic Events | From admission to discharge (up to 28 days) and at follow-up visits at 1 and 6 months post-surgery.
  Incidence of thrombotic events, including deep vein thrombosis, myocardial infarction, ischemic stroke, and pulmonary embolism.
Hyperkalemia | From the start of medication until 3 days after the end of treatment.
  Occurrence of elevated potassium levels (hyperkalemia) during the perioperative period.
Metabolic Acidosis | From the start of medication until 3 days after the end of treatment.
  Incidence of metabolic acidosis as measured by blood gas analysis.
Neurological Side Effects (Dizziness, Drowsiness, Seizures) | From the start of medication until 3 days after the end of treatment.
  Occurrence of neurological side effects, including dizziness, drowsiness, or seizures, reported by participants or physicians.
Gastrointestinal Side Effects | From the start of medication until 3 days after the end of treatment.
  Incidence of gastrointestinal side effects, including nausea, vomiting, indigestion, and diarrhea.
Limb Edema | From the start of medication until 3 days after the end of treatment.
  Occurrence of edema in the limbs during the medication period.
Upper Respiratory Tract Infections | From the start of medication until 3 days after the end of treatment.
  Incidence of upper respiratory tract infections during the medication period.
Allergic Reactions | From the start of medication until 3 days after the end of treatment.
  Occurrence of allergic reactions to the medication or other substances during the medication period.
Insomnia | From the start of medication until 3 days after the end of treatment.
  Incidence of insomnia reported by participants during the medication period.
Acute Kidney Injury | From the start of surgery until hospital discharge or within 4 weeks post-surgery.
  Incidence of acute kidney injury as defined by KDIGO criteria.
Postoperative Infections | From the start of surgery until hospital discharge or within 4 weeks post-surgery.
  Incidence of infections following surgery, including sepsis and pneumonia.
Mortality Rate | From the start of surgery until follow-up visits at 1 and 6 months post-surgery.
  All-cause mortality during the perioperative period and follow-up.
MACE (Major Adverse Cardiovascular Events) | From the start of surgery until follow-up visits at 1 and 6 months post-surgery.
  Incidence of MACE, including all-cause mortality, non-fatal myocardial infarction, and non-fatal stroke.
Other New Adverse Reactions | From admission to discharge (up to 28 days) and at follow-up visits at 1 and 6 months post-surgery.
  Any other newly reported adverse reactions that were not pre-specified but occurred during the perioperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, MD, PhD, Study Chair — Zhejiang University
Locations (1):
- Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No